CLINICAL TRIAL: NCT07298031
Title: How Can We Help? Wellbeing Interventions for Choral Music Ensembles
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jess Walls (Other)
Responsible Party: Sponsor-Investigator, Jess Walls, Principal Investigator, Auburn University
Organization: Auburn University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000298
Record Dates: First submitted 2025-12-11; First posted 2025-12-22 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Well-Being (Psychological Flourishing); Performance Anxiety
Keywords: Choral music; Wellbeing; Music; Anxiety; Performance anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: All study participants in the experimental group will receive the same interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Choral Interventions (Experimental): The interventions include box breathing, "Magnify", and emotion regulation through choral literature.
  Interventions: Behavioral: Box breathing; Behavioral: Magnify; Behavioral: Emotion regulation through choral literature

INTERVENTIONS:
Behavioral: Box breathing — Students will be led through a standard choral music breathing technique known as abdominal breathing, where they are reminded that a deep breath should cause your abdomen to expand to make more room in the lungs for air. After 2-3 standard deep breaths, they will be introduced to box breathing, which is an inhale for 4 beats, hold for 4 beats, exhale for 4 beats, hold for 4 beats, and repeat. Students will be told that this technique is useful for improving choral singing but can also be used in situations where the student is experiencing anxiety.
Behavioral: Magnify — This is a mindfulness-based technique that pulls from Cognitive Behavior Therapy and Dialectical Behavior Therapy techniques that is referred to colloquially as "what would happen if" or "magnify", used to examine cognitive distortions and reframe them to be more in line with reality. Students will be asked to think about an upcoming performance that may make them feel anxious and come up with a catastrophic scenario where everything that could possibly go wrong does go wrong, making note of the likelihood of the catastrophe. Students will internally come up with a best-case scenario and likelihood, and finally a most likely scenario somewhere between the best and worst case options.
Behavioral: Emotion regulation through choral literature — This intervention will use choral music literature to help students identify emotions, connect those emotions to their own experiences, and use the choral music literature to experience and work through those emotions in a safe environment. The choir will read through the lyrics of the chosen song, then narrow down the emotions referred to in the song using a list of possible emotions provided by the researcher. Students will recall an event in their own lives where they experienced that emotion, which they are not required to share out loud. With that emotion in mind, students will sing through the choral music piece, taking care to connect their own emotional experience with what they are singing. After the song, students will be asked to reflect on whether their own experiences with that emotion changed their perspective on the song, and whether singing about the emotion helped them work through their own situations and regulate their feelings.

SUMMARY:
The goal of this clinical trial is to learn if psychology and music based interventions can impact anxiety and overall wellbeing in adolescents enrolled in choral music classes. The main questions it aims to answer are:

Do specific psychology and music based breathing interventions impact anxiety and overall wellbeing in adolescents? Do specific psychology and music based performance anxiety reduction interventions impact anxiety and overall wellbeing in adolescents? Do specific psychology and music based emotion regulation interventions impact anxiety and overall wellbeing in adolescents? Researchers will compare results of pre-test data, post-test data, qualitative interviews, and surveys of adult choral directors to see if there is a measurable impact on adolescent anxiety and overall wellbeing.

Participants will:

* Use box breathing during choral music warm-ups to connect choral breathing to breathing for anxiety reduction
* Use "magnify" technique to compare cognitive distortions regarding an upcoming performance that may cause anxiety to the most likely realistic outcome
* Use emotion regulation through song lyrics technique to connect lyrics of choral music repertoire to participants experienced emotions

DETAILED DESCRIPTION:
The research design is experimental mixed-methods, designed to determine the effectiveness of specific breathing and mindfulness techniques and specific emotion regulation techniques. These techniques are hypothesized to be useful in reducing anxiety and improving overall emotion regulation and wellbeing when integrated into choral music ensemble rehearsal practices, with additional determinations made regarding the effectiveness of these techniques in improving the quality of musical performance. This project incorporates techniques many music educators already employ, but with a better understanding of the psychology involved and specific wellbeing goals, to measure the effectiveness of these interventions and provide both evidence of effectiveness and a standard way to provide training on these interventions to music educators.

Participants are middle school and high school students in grades 6 through 12 who are currently enrolled in a choir class in Fort Bend ISD, Texas. One high school and one middle school campus will serve as a control group, with that group only taking the pre-test and receiving no interventions, and a second high school and middle school will serve as the primary experimental study sites. Individual schools were chosen due to administration and choral music educators who support educational research, with the experimental school sites and control school sites as closely matched demographically as possible, with all 4 sites having strong choral music programs. The experimental middle school is the experimental high school feeder, and the control middle school is the control high school feeder.

The instrument for the initial pre-test survey includes 21 items on a 4-point Likert scale ranging from "A bit like me" to "A lot like me" in three categories: Emotion, Music and Emotions, and Music and Anxiety, along with basic demographic information. Student information was anonymized by identifying individuals exclusively by choir folder number, to correlate pre- and post-test data. Example survey items include "I know what to do when I feel a difficult emotion." and "I have had a strong emotional reaction to one or more songs we have performed or sung in choir." This 21-item rating scale was pilot tested in an educational methods survey design course. The pre-test survey also included questions from the GAD-7, WEMWBS, and DERS-SF. The pre-test survey will be administered to both the control group and the experimental group.

The post-test survey contains all questions from the pre-test survey, with an additional five rating scale questions and one open-ended question for participants to add information regarding anxiety, positive emotions, emotion regulation, and the intervention techniques in their own words. This survey will be given only to the experimental group and will be administered twice: once immediately after the intervention, and once a week later.

Participants and their parents will self-identify willingness to participate in a follow-up interview on the consent/assent form, with two to three participants per class period selected at random by folder number from the self-identified willing participants. These interviews will be scheduled at the end of the initial research administration day to occur one week later at the follow up, will be approximately 15-20 minutes long, and will be conducted immediately after the second administration of the post-test. The parents of the minor participants will be invited to join the interview either via zoom or in person and have the option of their choir director attending the interview in their place. Parents and participants can opt out of the interview at any time with no penalties, with one or two extra participants selected on a stand by basis per class in case of absence or the choice to opt out of the interview.

Choir directors will participate in a follow-up survey approximately one month after the initial intervention, which includes 12 open-ended questions for the director to answer on their own time. This survey will be on Qualtrics, and will be distributed to the three participating choir directors by email approximately four weeks after the initial intervention, with a request to complete the survey within one calendar week. A follow-up email will be sent five days after the survey was distributed to any directors who had not yet completed the survey.

A timeline of study activities for intervention groups:

Prior to interventions:

* All students given pre-test survey online on Qualtrics Intervention 1: Box Breathing
* Students will be led through standard choral music abdominal breathing, placing hands between rib cage and hip bones to ensure deep inhalation is taking place. Students will take 2-3 of these deep breaths.
* Students will be taken through box breathing

  * "Class, now I am going to take you through something called box breathing. If you have not heard of it, that's ok, it's a pretty easy thing to learn as long as you can count to 4. As a reminder, if at any point this is too stressful or you feel the need to sit out, you are welcome to take a seat, ask your choir director for permission to leave the room, or even ask for a pass to the counselor if you are feeling really anxious. First, you take a deep abdominal breath like we just practiced for a count of 4, try it with me, 1-2-3-4. Now, hold with that breath in for a count of 4, 1-2-3-4. Now, slowly exhale for 4, 1-2-3-4. Last, hold with that breath exhaled, 1-2-3-4. Ok, now that we know how that goes, we are going to practice it a few times, in-2-3-4, hold-2-3-4, out-2-3-4, hold-2-3-4. One more time, in-2-3-4, hold-2-3-4, out-2-3-4, hold 2-3-4."
  * "Ok, now here is the part that is a little different than your normal choir breathing. This particular type of breathing is not just good for singing, it is also really helpful for anxiety. If you're not familiar with anxiety, that's when you're stressed out or scared about something to the point that it might make you feel a little sick, and it's really hard to get that thing out of your head. It happens to pretty much everyone at some point, and it's not fun, but there are some really good ways you can help your body regulate when you're feeling anxious, and box breathing is one of them. So this time, when we do the box breathing, I want you to think of something that has been stressing you out. Maybe don't pick something really big and stressful, pick something kind of mid-level stressful, like worrying about a test coming up next period."
  * Take a pause. "Ok, do you have your mid-level stressful thing in mind? With that thing in mind, let's do three rounds of box breathing. Ready, in-2-3-4, hold-2-3-4, out-2-3-4, hold-2-3-4. Again, in-2-3-4, hold-2-3-4, out-2-3-4, hold-2-3-4. One more time, in-2-3-4, hold-2-3-4, out-2-3-4, hold-2-3-4. Hopefully that helped you feel a little better, a little more regulated, it might take some practice for it to help, so try it when you have little things in your life that stress you out. When your mom tells you to clean your room when you're in the middle of doing your homework and you just want to explode, try box breathing first and see if that helps you be a little calmer when you address the situation." Intervention 2: "Magnify" technique.
* Students will go through a scenario thinking about their next upcoming performance, first imagining everything that could possibly go wrong, then imagining the best possible outcome, then brainstorming the most likely outcome.

  * "Ok, this one may be a little different. You don't have to raise your hand, but are any of you nervous about performing? You get up on stage, and get a bit of stage fright or anxiety and maybe feel butterflies in your stomach or feel like you might throw up? That is a really normal thing, and I want to try something to see if we can help reduce some of that anxiety about performing. Just like before, if at any point this is too stressful or you feel the need to sit out, you are welcome to take a seat, ask your choir director for permission to leave the room, or even ask for a pass to the counselor if you are feeling really anxious. This one might stress you out just a little at first, but if you stick with me, I think it will really help make performing feel a little less scary."
  * "First, I want you to think of your upcoming performance. It is at [location], on [date]. One of the most stressful parts of a performance is worrying that something will go wrong, so I want you to take a moment and imagine absolutely everything that could possibly go wrong. It's ok if those thoughts are both totally reasonable things like you start to sing and have a frog in your throat and it's really loud (happened to me during my first solo), or your piano player drops their music and stops playing (happened to me in college), or it can be rather absurd things like a light crashing down on the stage. Whatever your brain wants to worry about with the most horrible things that could happen, let it worry for just a minute, without judging yourself for thinking something silly."
  * "Now that you've thought of all of those terrible things that can happen, I want you to put all of those terrible things in a box for a moment, and set them to the side. We're going to think about the best possible outcome now. If absolutely everything went the best it possibly could at this performance, what would that look like? Think about things like everyone coming up to you afterward and saying your performance was incredible, gave them goosebumps, made them cry. Think about your family and friends offering to buy you ice cream, or giving you flowers or presents because it was so amazing. You can let these thoughts get a little absurd too, think about if Taylor Swift was somehow at the concert and asked your choir to come perform at the Eras tour. Again, don't judge yourself and let it be a little silly."
  * "Next, I want you to take back out that box of terrible things, and put your box of wonderful things next to it. Think about your terrible things one by one, and try to consider how likely they are to happen. Getting a frog in your throat is probably the most likely to happen, like I said it did happen to me on my very first solo ever. Since that day, I have performed hundreds of times, and it has never happened again, so that is what, maybe at most a 1 in 100 chance? So it's possible, but is it really likely? And even if it happens, is it going to ruin the rest of the performance? Not if you are prepared to keep going no matter what happens, after that a few people noticed, but most people congratulated me on doing a fantastic job after that rough start, they didn't focus on the mistake but on how I came back from it. Same story with the piano player dropping his music, I kept singing, he came back in, and I was praised for continuing on despite things getting tricky. And again, that was maybe at most a 1 in 100 chance of happening. Some slightly more common things that could happen are someone locking their knees and passing out during a performance, but even that is probably a 1 in 25 or maybe 1 in 50 chance, and when it does happen, the people around them usually step in to help catch them and help them sit down, and the performance continues. If something catastrophic happens, which by my estimates is at most a 1 in 1,000 chance, your director will be the one to take charge, and one of the most beautiful things in the world is people coming together to help other people when something bad happens. You might be thinking, what if we just sing really badly? Well, that could happen, but you've prepared for this moment, you've worked really hard, you have a great director. Even if it happens, you chalk that up to a learning opportunity and make sure you practice more next time so it won't happen again."
  * "Last, let's think about the most likely scenario for this performance. You probably won't be invited to a Taylor Swift performance, but you also probably won't be booed off the stage. The most likely scenario is that you will sing and perform your very best, maybe with a small mistake or two, and your families and friends in the audience will be really proud of you. Those little mistakes will be something you can learn from, and do better next time you have a performance, because without making mistakes we don't really have anything to learn from. Next time you have a performance, try thinking through it like this, first the worst that could happen, then the best, then the most likely, and see if that helps you feel a little less anxious, because even if things aren't perfect, they will still more than likely be pretty good, and even if they're not you will learn from them." Intervention 3: Emotion Regulation using Choral Music Literature
* Students will open their music to a selected song from their current music repertoire.

  * "Looking at this song, let's read the lyrics together." Read lyrics, with emotional conviction. "Listening to those lyrics, what general emotion comes to mind? Looking at this chart (provided below in this document), which of the main emotions seems to fit best between Happy, Sad, Angry, Afraid, and Ashamed? Ok, looking at the emotion we chose, would you say this song is high intensity, medium intensity, or low intensity? Which of the emotions within that category seems to fit this song the best?" Read off the emotions in the selected category, there may be a few that fit, we will stick with the one that receives the most consensus from the group. This will differ in every song.
  * "Ok, now that we have narrowed down what the main emotion is in this song, I want you to think about a time in your own life that you have felt that emotion. You do not have to share that experience out loud, it is only for you. Think about what happened that caused you to feel that emotion, and how you reacted in the moment to that emotion. Think about whether your reaction to that emotion matched the situation, or if maybe you reacted with more or less intensity than the situation may have called for. For example, if the emotion was sad, and I thought about a time I wanted cereal for breakfast, but I went to the cupboard and my son had eaten the last of the cereal, and I felt so sad that I sat down on the floor in the kitchen and cried my eyes out, that is me feeling the correct emotion, but maybe at an intensity level that didn't quite fit the situation. On the other hand, if the emotion was happy and I just found out I won a million dollars, and I just said 'oh that's nice' and went on with my day, again that is the right emotion but too low of an intensity for the situation. It's not necessarily a bad or good thing to react to your emotions with the wrong intensity, just something to be aware of and see if you can figure out why your reactions don't quite match."
  * "Going back to your experience with the emotion we just named for this song, I want you to read the words to yourself silently, picturing that experience you had with this emotion while you read the words. See if you can make a deeper emotional connection to the song by thinking about your own life, and connecting to what the words really mean. Now, with that connection in mind, we are going to sing through the song all together. We are not going to worry as much about right or wrong notes, we are just focusing on singing this song with a deeper connection to the emotion because of our own experiences. While we are doing that, I want you to think about letting the song be your expression of that emotion, so you can let go of it if you feel like you need to."
* Students will then sing through the song, focusing on their own emotional experience. I will not ask them to share what that was like for them, as that will be part of the post-test they will take.

After intervention:

• One week after the intervention, the researcher will return, give the final post-test, and conduct interviews with members of the experimental group.

Quantitative data will be analyzed using descriptive statistics and mixed ANOVA using SPSS software, comparing data for individual students within the intervention group, and comparing pre-test data for the control group to the data from the intervention group. Qualitative data from interviews and the open-ended choir director survey will be coded inductively by the researcher and a research methodologist from the dissertation committee.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in 6th through 12th grade at selected schools
* Enrolled in choir at the selected schools

Exclusion Criteria:

* None

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety | From enrollment to choir director survey 4 weeks later
  Measured quantitatively through:
  -pre-test and post-test data
  Measured qualitatively through:
  * Student interview questions exploring experiences of anxiety and use of breathing and "Magnify" techniques
  * Qualitative responses to open-ended post-test survey items
  * Choir director observations of anxiety and performance anxiety (open-ended director survey)
Change in Emotion Regulation | From enrollment to the choir director survey 4 weeks post intervention
  Measured quantitatively through:
  -pre-test and post-test data
  Measured qualitatively through:
  * Student interview questions exploring emotional processing during the music-based intervention
  * Post-test open-ended responses regarding emotion regulation
  * Choir director survey reporting observed changes in students' emotion regulation
Change in Well-Being | From enrollment to second post-test administration one week after intervention
  Measured quantitatively through:
  -pre-test and post-test data
  Measured qualitatively through:
  * Interview comments about perceived overall well-being changes
  * Open-ended post-test items about intervention effectiveness

SECONDARY OUTCOMES:
Change in Musicality and Emotional Engagement in Music | From enrollment to choir director survey 4 weeks after intervention
  Measured qualitatively through:
  * Choir director open-ended survey addressing musicality, emotional expression, and performance anxiety
  * Qualitative coding of director observations and researcher field notes
  Measured indirectly through:
  -Student reflections on connecting emotion to choral literature in interviews and post-test items

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kuehne, PhD, Study Chair — Auburn University
Locations (1):
- Fort Bend ISD, Sugar Land, Texas, United States

IPD SHARING:
Plan to Share IPD: No